CLINICAL TRIAL: NCT07008391
Title: High-Sensitivity Troponin I in Addition to Guideline-Based Care in Emergency Medical Service - an Open Randomized Controlled Trial
Brief Title: High-Sensitivity Troponin I in Addition to Guideline-Based Care in EMS
Acronym: TIGER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Ambulance care in Greater Stockholm Ltd (AISAB), Region Stockholm (Unknown)
Responsible Party: Principal Investigator, Jakob Lederman, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-07919-01
Record Dates: First submitted 2025-05-16; First posted 2025-06-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Emergency Medical Services; Nursing Care; Cardiology; Myocardial Infarction; Myocardial Infarction or Chest Pain; Myocardial Infarction, Acute; Emergencies; Ambulance
Keywords: Ambulance; Prehospital emergency nurse; Sweden; Point-of-care; troponin; high sensitive troponin
MeSH Terms: conditions — Myocardial Infarction; Chest Pain; Emergencies

STUDY DESIGN:
Intervention Model Description: 2:1 Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Getting a point-of-care Troponin I analysed, in addition to care according to medical guidelines in EMS
  Interventions: Diagnostic Test: high sensitivity Troponin I
- Control (No Intervention): Getting care according to medical guidelines in EMS

INTERVENTIONS:
Diagnostic Test: high sensitivity Troponin I — Study participants in the intervention group will have the high-sensitivity Troponin I blood test analyzed during emergency medical service (EMS) care using the point-of-care Siemens Atellica® VTLi system. The test result will be documented in the EMS electronic medical record (FRAPP), transmitted along with the ECG, and communicated verbally to the receiving hospital during handover.
  Arms: Intervention

SUMMARY:
The TIGER study is a study investigating the utlility of a point-of-care blood analyse of Troponin I to help identify patients with heart attacks in the prehospital emergency care. The study is conducted within the ambulance services of Region Stockholm and compares standard medical care with and without the addition of this quick test.

Chest pain is one of the most common reasons for ambulance dispatch, but currently only about one-third of heart attacks are detected before arriving at the hospital-mainly through ECG. The remaining two-thirds are not identified until after further testing at the emergency department. The TIGER study aims to improve early diagnosis by using a high-sensitivity, point-of-care Troponin I test already in the prehospital phase.

The study is a randomized controlled trial, where participants are randomly assigned to one of two groups. One group receives standard emergency care along with the rapid Troponin I test in the ambulance. The other group receives standard care without the test. The goal is to evaluate whether the use of Troponin I testing leads to faster and more accurate identification of heart attacks, ultimately improving patient outcomes.

In total, about 1,419 adult patients with chest pain or suspected heart attack will participate. The primary outcome being measured is the time from first medical contact to PCI (balloon angioplasty). Secondary outcomes include time spent in different parts of care, hospital length of stay, the occurrence of serious events (such as heart attack, stroke, or death), and the diagnostic accuracy of the test.

The study has been approved by the Swedish Ethical Review Authority and includes safety monitoring through an interim analysis after the first 150 patients. Test results from the Troponin I analysis are clearly marked as part of the research study and should be interpreted by the responsible physician alongside other clinical findings.

DETAILED DESCRIPTION:
The TIGER study is a prospective, open-label, randomized controlled trial designed to evaluate the clinical utility of prehospital high-sensitivity Troponin I testing in patients presenting with chest pain or suspected myocardial infarction (MI). The study is conducted within the emergency medical services (EMS) in Stockholm, Sweden.

Participants are randomized in a 2:1 ratio to receive either standard guideline-based care alone or standard care plus point-of-care Troponin I testing using the Siemens Atellica® VTLi system. The Troponin result is available to EMS providers in real-time and is communicated to the receiving hospital as part of the routine prehospital handover.

The study aims to assess whether the addition of early biomarker data can improve triage, reduce time to treatment (FMC-to-balloon time), and optimize the use of healthcare resources. An interim analysis will be conducted after 150 patients have been enrolled. The study has been approved by the Swedish Ethical Review Authority.

ELIGIBILITY:
Inclusion Criteria:

* Chestpain / discomfort and/or
* Clinical suspicion of myocardial infarction by the prehospital personeel

Exclusion Criteria:

* Patients suffering from a trauma and conveyed to the trauma level 1 hospital.
* Missing valid social security number
* Not beeing able to give informed consent
* Not a primary assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1419 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Time from First Medical Contact to Vascular Access (FMC-to-Access Time) | From time of first medical contact by EMS to time of vascular access during index PCI procedure, assessed during index hospitalization (typically within 72 hours)
  Time in minutes from the initial contact with emergency medical services (EMS) to vascular access (arterial puncture) for percutaneous coronary intervention (PCI), representing the time to initiation of the invasive procedure.

SECONDARY OUTCOMES:
Time from First Medical Contact to Initial ECG (FMC-to-ECG Time) | From time of initial patient contact by EMS personnel to time of first ECG, assessed during prehospital phase (typically within 1 hour)
  Time in minutes from the first contact with emergency medical services (EMS) personnel-defined as the moment EMS arrives at the patient-to completion of the first 12-lead ECG.
Time from First Medical Contact to Emergency Department Admission (FMC-to-ED Admission Time) | From time of first medical contact to ED admission, assessed on the day of presentation (typically within 4 hours)
  Time in minutes from first EMS contact to arrival and registration at the emergency department.
Emergency Department Length of Stay | From time of ED admission to ED discharge, assessed during index visit (typically within 24 hours)
  Duration in minutes from emergency department registration to transfer or discharge from the ED.
Total Hospital Length of Stay | From ED admission to hospital discharge, assessed during index hospitalization (up to 14 days)
  Duration in minutes from emergency department admission to hospital discharge (from acute care facility).
Major Adverse Cardiovascular Events (MACE) | Assessed at 72 hours and at 30 days from the time of first medical contact, defined as the arrival of emergency medical services (EMS)
  Composite outcome including the occurrence of any of the following within the specified time frames: myocardial infarction, angina pectoris, all-cause mortality, stroke, or heart failure with reduced ejection fraction (HFrEF).
Number of Interventions Performed During Acute Care Episode | From the time of first medical contact-defined as the arrival of EMS personnel at the patient's side-through hospital discharge, assessed during the full acute care episode (up to 14 days)
  Total number of interventions performed per patient from first medical contact through hospital discharge. Interventions may include prehospital treatments (e.g., defibrillation, medication administration) and in-hospital procedures such as diagnostic angiography, percutaneous coronary intervention (PCI), temporary pacing, or surgery.
Proportion of participants assigned to in-hospital care | From admission to discharge, during index hospitalization (up to 14 days)
  Proportion of participants assigned to each predefined category of in-hospital care, based on the most resource-intensive setting they were treated in during the index hospitalization. The categories include:
  * Emergency Department (ED) only
  * Direct to Percutaneous Coronary Intervention (PCI)
  * Cardiac Intensive Care Unit (CICU)
  * Intermediate Care Unit
  * Other Cardiac Unit
  * General Care Unit
  * External Care Institution (e.g., step-down or rehabilitation facility)
  Unit of Measure: Percentage of participants (%)
Clinical Utility: Sensitivity, Specificity, Negative Predictive Value (NPV), and Positive Predictive Value (PPV). | From the time of EMS assessment (first medical contact) to confirmation of final diagnosis at hospital discharge (typically within 7-14 days)
  Diagnostic performance of prehospital assessment for identifying patients with Myocardial infarction. Includes calculation of sensitivity, specificity, negative predictive value (NPV), and positive predictive value (PPV), using confirmed diagnosis (ICD-code) at discharge as reference standard.
Incidence of Other Time-Critical Medical Conditions | Assessed up to 30 days from the time of first medical contact by emergency medical services (EMS)
  Number of participants diagnosed with other time-critical medical conditions within 30 days of first medical contact. These may include but are not limited to: stroke, sepsis, aortic dissection, pulmonary embolism, or major trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Lederman, PhD, Principal Investigator — Karolinska Institute, Department of Clinical Science and Education; Veronica Vicente, Docent, Study Chair — Karolinska Institute, Department of Clinical Science and Education
Locations (1):
- Ambulance care in greater Stockholm Ltd. (AISAB), Stockholm, Årsta, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because consent for data sharing was not obtained from participants and data sharing is not feasible due to ethical restrictions

DOCUMENTS (3):
  • Study Protocol (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT07008391/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT07008391/SAP_001.pdf
  • Informed Consent Form (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT07008391/ICF_002.pdf